CLINICAL TRIAL: NCT03247192
Title: Effect of Whey Protein Supplementation Associated With Resistance Training on Body Composition, Cellular Hydration, Phase Angle, Muscle Strength, Glycemic and Lipid Profile, Inflammatory and Oxidative Stress Markers in Trained Older Women
Brief Title: Whey Protein Supplementation Associated With Resistance Training on Health Indicators in Trained Older Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Collaborators: Coordination for the Improvement of Higher Education Personnel (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Hellen Clair Garcêz Nabuco, master degree, Universidade Estadual de Londrina
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: UEL1700756-1/2016
Record Dates: First submitted 2017-08-08; First posted 2017-08-11 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Body Composition; Healthy
Keywords: resistance training; protein supplementation; aging; Randomized Controlled Trial
MeSH Terms: interventions — Placebo Effect

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (3):
- Whey protein-placebo (Experimental): Participants received a dose of 35 grams of whey protein before resistance training (RT) and a dose of 35 grams of maltodextrin (placebo) after RT.
  Participants were personally supervised by physical education professionals with substantial RT experience. The sessions were performed 3 times per week on Mondays, Wednesdays, and Fridays, with 3 sets of 08-12 repetition maximums. The RT program was a whole-body program with eight exercises, including: chest press, seated row, triceps pushdown, preacher curl, horizontal leg press, knee extension, leg curl and seated calf raise. Participants were afforded a 1 to 2 min rest interval between sets and 2 to 3 min between each exercise. The training load was consistent with the prescribed number of repetitions for the three sets of each exercise.
  Interventions: Dietary Supplement: Whey protein-placebo
- Placebo-whey protein (Experimental): Participants received a dose of 35 grams of maltodextrin (placebo) before resistance training (RT) and a dose of 35 grams of whey protein after RT.
  Participants were personally supervised by physical education professionals with substantial RT experience. The sessions were performed 3 times per week on Mondays, Wednesdays, and Fridays, with 3 sets of 08-12 repetition maximums. The RT program was a whole-body program with eight exercises, including: chest press, seated row, triceps pushdown, preacher curl, horizontal leg press, knee extension, leg curl and seated calf raise. Participants were afforded a 1 to 2 min rest interval between sets and 2 to 3 min between each exercise. The training load was consistent with the prescribed number of repetitions for the three sets of each exercise.
  Interventions: Dietary Supplement: Placebo-whey protein
- Placebo-placebo (Placebo Comparator): Participants received a dose of 35 grams of maltodextrin (placebo) before and after resistance training.
  Participants were personally supervised by physical education professionals with substantial RT experience. The sessions were performed 3 times per week on Mondays, Wednesdays, and Fridays, with 3 sets of 08-12 repetition maximums. The RT program was a whole-body program with eight exercises, including: chest press, seated row, triceps pushdown, preacher curl, horizontal leg press, knee extension, leg curl and seated calf raise. Participants were afforded a 1 to 2 min rest interval between sets and 2 to 3 min between each exercise. The training load was consistent with the prescribed number of repetitions for the three sets of each exercise.
  Interventions: Dietary Supplement: Placebo-placebo

INTERVENTIONS:
Dietary Supplement: Whey protein-placebo — This investigation was carried out over a period of 26 weeks divided in two phases. The first phase of the study was an eight-week period (weeks 3-10), during which subjects were familiarized to RT. Phase 2, supplementation phase, the participants was randomized in three groups and started 12 weeks dedicated to supplementation plus RT (weeks 13-24). At the beginning and the end of each phase of the experiment, two weeks were allocated for evaluations (weeks 1-2, 11-12 and 25-26) consisting of anthropometric, body composition, blood samples, blood pressure, one repetition maximum tests (1RM) and dietary intake measurements
  Arms: Whey protein-placebo
Dietary Supplement: Placebo-whey protein — This investigation was carried out over a period of 26 weeks divided in two phases. The first phase of the study was an eight-week period (weeks 3-10), during which subjects were familiarized to RT. Phase 2, supplementation phase, the participants was randomized in three groups and started 12 weeks dedicated to supplementation plus RT (weeks 13-24). At the beginning and the end of each phase of the experiment, two weeks were allocated for evaluations (weeks 1-2, 11-12 and 25-26) consisting of anthropometric, body composition, blood samples, blood pressure, one repetition maximum tests (1RM) and dietary intake measurements
  Arms: Placebo-whey protein
Dietary Supplement: Placebo-placebo — This investigation was carried out over a period of 26 weeks divided in two phases. The first phase of the study was an eight-week period (weeks 3-10), during which subjects were familiarized to RT. Phase 2, supplementation phase, the participants was randomized in three groups and started 12 weeks dedicated to supplementation plus RT (weeks 13-24). At the beginning and the end of each phase of the experiment, two weeks were allocated for evaluations (weeks 1-2, 11-12 and 25-26) consisting of anthropometric, body composition, blood samples, blood pressure, one repetition maximum tests (1RM) and dietary intake measurements
  Arms: Placebo-placebo

SUMMARY:
The main purpose of the present study was to investigate the effects of whey protein supplementation associated with resistance training on muscle strength, body composition, muscle quality, cellular hydration, cardiometabolic risk factors, inflammatory and oxidative stress markers in trained elderly women and to evaluate whether the timing of protein intake provide different responses on these variables.

DETAILED DESCRIPTION:
This study was carried out over a period of 26 weeks divided in two phases. The first phase of the study was an eight-week period (weeks 3-10), during which subjects were familiarized to RT. This RT period was conducted to standardize training status, and to overcome strong neural adaptations known to occur within the first few weeks of RT. Phase 2, supplementation phase, the participants was randomized in three groups and started 12 weeks dedicated to supplementation plus RT (weeks 13-24). At the beginning and the end of each phase of the experiment, two weeks were allocated for evaluations (weeks 1-2, 11-12 and 25-26) consisting of anthropometric, body composition, one repetition maximum tests (1RM), phase angle, body water, blood samples and dietary intake measurements.

Recruitment was carried out through newspaper and radio advertising, and home delivery of leaflets in the central area and residential neighborhoods. All participants completed health history and physical activity questionnaires and met the following inclusion criteria: 60 years old or more, physically independent, free from cardiac or orthopedic dysfunction, not receiving hormonal replacement and/or thyroid therapy, not using equipment that would prevent the accomplishment of protocols and tests, and not performing any regular physical exercise for 6 months preceding the beginning of the study. Participants have passed a diagnostic graded exercise stress test with 12-lead electrocardiogram reviewed by a cardiologist and were released with no restrictions for participation in this investigation. Eighty-three Brazilian older women (≥ 60 years old), volunteered to participate in this investigation. After individual interviews, thirteen volunteers were excluded because they did not meet the inclusion criteria. Seventy participants were submitted to a standardized resistance training (RT) program, for eight weeks. After the assessments, the participants were randomly divided into three groups according relative strength (ratio of total strength obtained on 1-RM tests by body mass): (1) whey protein pre- and placebo post- RT (whey protein-placebo, (2) placebo pre- and whey protein post- RT, and (3) placebo pre- and post- RT. A blinded researcher was responsible for generating random numbers for participant allocation. All groups were submitted to the same RT program and 66 participants completed the experiment. The reasons for withdrawal from the study was reported as personal reasons and transportation issues.

Written informed consent was obtained from all participants after a detailed description of investigation procedures was provided. This investigation was conducted according to the Declaration of Helsinki and was approved by the local University Ethics Committee (nº 1.700.756).

The paired t-test was used to analyze the effects (pre- vs post-) of the first phase. Two-way analysis of variance for repeated measures was applied for intra- and inter-group comparisons. When the baseline was different (ANOVA one-way), two-way analysis of covariance (ANCOVA) for repeated measures was applied for comparisons, with baseline scores used as covariates. When an F-ratio was significant, Fisher's post hoc test was employed to identify mean differences. The statistical power was determined to verify the statistical power of the analysis. For all statistical analyses, significance was accepted at P<0.05.

ELIGIBILITY:
Inclusion Criteria:

* 60 years old or more, physically independent, free from cardiac or orthopedic dysfunction, not receiving hormonal replacement therapy, and not performing any regular physical exercise more than once a week in the six months preceding the beginning of the investigation
* Participants passed a diagnostic graded exercise stress test with a 12-lead electrocardiogram, reviewed by a cardiologist, and were released with no restrictions for participation in this investigation.

Exclusion Criteria:

* All subjects not participating in 85% of the total sessions of training or withdraw

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-12-08; Primary Completion 2016-02-10 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Change in body composition | baseline 1; after 8 weeks (baseline2) and after 12 weeks
  Whole-body dual-energy X-ray absorptiometry (DXA) (Lunar Prodigy) was used to assess lean mass and fat mass and its segments. The total skeletal muscle mass (SMM) was estimated by the predictive equation proposed by Kim et al. (Kim et al., 2004). The results are presented in kg.
Change in Phase Angle | baseline 1; after 8 weeks (baseline2) and after 12 weeks
  Spectral bioelectrical impedance device (Xitron Hydra, model 4200, San Diego, CA, USA) was used to estimate the resistance (R), and reactance (Xc), and subsequently the phase angle (PhA) was calculated as arc-tangent (Xc/R) x 180°/π. The results are presented in degree
Change in cellular hydration | baseline 1; after 8 weeks (baseline2) and after 12 weeks
  Spectral bioelectrical impedance device (Xitron Hydra, model 4200, Xitron Technologies, San Diego, CA, USA) was used to estimate the intracellular water (ICW), extracellular water (ECW), and total body water (TBW). The results are presented in liters (L)
Change in C-reactive protein (CRP) | baseline 1; after 8 weeks (baseline2) and after 12 weeks
  Measurements of serum levels of high-sensitivity CRP were carried out using a biochemical auto-analyzer system (Dimension Max - Siemens Dade Behring) according to established methods in the literature consistent with the manufacturer's recommendations. The results are presented in milligrams per decilitre (mg/dL).
Change in inflammatory markers | Baseline and 12 weeks
  Tumor Necrosis Factor -α (TNF-α) and Interleukin-6 (IL-6) were determined by enzyme-linked immunosorbent assay (ELISA), according to the specifications of the manufacturer (Quantikine High Sensitivity Kit, Minneapolis) and performed in a microplate reader Perkin Elmer, model EnSpire (Waltham, MA, USA). All samples were determined in duplicate to guarantee the precision of the results. The results are presented in picograms per milliliter (pg/ml).
Change in CATALASE (CAT) | Baseline and 12 weeks
  The CAT analysis is by measuring the decay in concentration of hydrogen peroxide
  , and oxygen generation using the technique described by literature. The reading of the CAT reaction was carried out in a spectrophotometer, ThermoSpectronic® brand, model HELIOS-α (Waltham, MA, USA) at a wavelength of 240 nm.
Change in superoxide dismutase (SOD) | Baseline and 12 weeks
  The SOD activity in erythrocytes was determined using the pyrogallol method described by literature. The reading of SOD reaction is performed in a spectrophotometer, thermoSpectronic® brand, model HELIOS-α (Waltham, MA, USA) at a wavelength of 420 nm.
Change in oxidative stress | baseline 1; after 8 weeks (baseline2) and after 12 weeks
  For measurements, advanced oxidation protein products (AOPP) were determined in the plasma using a semiautomatic method. AOPP concentrations were expressed as micromoles per liter (μmol/L). Total plasma antioxidant capacity (TRAP) was determined by the chemiluminescence method for the induction time of 2.2 azo-bis (2-amidinopropane) and calibrated with Trolox analogue of vitamin E. TRAP values were expressed in μmol of Trolox.
Change in lipid profile | baseline 1; after 8 weeks (baseline2) and after 12 weeks
  Measurements of serum levels of total cholesterol (TC), high-density lipoprotein (HDL-C) and triglycerides (TG) were determined using a biochemical auto-analyzer system (Dimension Max - Siemens Dade Behring) according to established methods in the literature consistent with the manufacturer's recommendations. For the determination of LDL-c was used the Friedewald equation: LDL-c=TC - (HDL-c + TG / 5). The Castelli Index I was calculated by dividing the total cholesterol concentration (TC) by the concentration of HDL-c (CT / HDL-c), while the Castelli Index II was determined from concentration of LDL-c divided by the concentration of HDL-c (LDL-c / HDL-c)
Change in glucose, insulin and HOMA-IR | baseline 1; after 8 weeks (baseline2) and after 12 weeks
  Measurements of serum levels of glucose (GLU) were determined using a biochemical auto-analyzer system (Dimension Max - Siemens Dade Behring).Insulin was determined by the chemiluminescence method (LIASON equipment) and the Homeostasis Assessment Model (HOMA-IR) was calculated by the formula: Insulin fasting (μUI / mL) x Glucose fasting (mmol / L) / 22.5.
change in Muscular strength | baseline 1; after 8 weeks (baseline2) and after 12 weeks
  Maximal dynamic strength was evaluated using the 1RM test assessed on chest press, knee extension, and preacher curl exercises performed in this exact order. Testing for each exercise was preceded by a warm-up set (6-10 repetitions), with approximately 50% of the estimated load used in the first attempt of the 1RM. This warm-up was also used to familiarize the subjects with the testing equipment and lifting technique. The testing procedure was initiated 2 minutes after the warm-up. The subjects were instructed to try to accomplish two repetitions with the imposed load in three attempts in both exercises. The rest period was 3 to 5 min between each attempt, and 5 min between exercises. The 1RM was recorded as the last resistance lifted in which the subject was able to complete only one single maximal execution

SECONDARY OUTCOMES:
Change in anthropometric measurements | baseline 1; after 8 weeks (baseline2) and after 12 weeks
  Body mass was measured to the nearest 0.1 kg using a calibrated electronic scale scale (Balmak), with subjects wearing light workout clothing and no shoes. Height was measured using a stadiometer to the nearest 0.1 cm while subjects were standing without shoes. Body mass index was calculated as the body mass in kilograms divided by the square of the height in meters. We also collected data on waist circumference (WC) and (HC) hip, using a flexible and inelastic tape measure. WC was obtained at the midpoint between the last rib and the iliac crest at the time of expiration and the WC was measured in the region of greater perimeter between the waist and the thigh. Two measurements were used to measure each circumference. In situations in which the difference between the measurements was greater than 0.5 cm a third measurement was performed, with the value of the median being adopted as reference. All measurements were performed by the same evaluator.
Change in blood pressure | baseline 1; after 8 weeks (baseline2) and after 12 weeks
  Resting BP assessment was performed using automatic, oscillometric equipment (Omron - 7113). Participants attended the laboratory on three different days and, during each visit, remained seated at rest for 10 min with the cuff of the equipment in place on the right arm. Subsequently, several BP measurements were performed at one-minute intervals in order to obtain three consecutive measurements where the difference in systolic BP (SBP) and diastolic BP (DBP) readings differed by no more than 4 mmHg. The average of the three measurements for each day was averaged across the three visits.
Dietary intake | baseline 1; after 8 weeks (baseline2) and after 12 weeks
  Food consumption were assessed by the 24-hour dietary recall method applied on two non-consecutive days of the week, with the aid of a photographic record taken during an interview. The homemade measurements of the nutritional values of food and supplementation were converted into grams and milliliters by the online software Virtual Nutri Plus (Keeple®, Rio de Janeiro, Rio de Janeiro, Brazil) for diet analysis. Some foods were not found in the program database and therefore items were added from food tables.

REFERENCES:
- [Background] American College of Sports Medicine. American College of Sports Medicine position stand. Progression models in resistance training for healthy adults. Med Sci Sports Exerc. 2009 Mar;41(3):687-708. doi: 10.1249/MSS.0b013e3181915670. PMID 19204579
- [Background] Kim J, Heshka S, Gallagher D, Kotler DP, Mayer L, Albu J, Shen W, Freda PU, Heymsfield SB. Intermuscular adipose tissue-free skeletal muscle mass: estimation by dual-energy X-ray absorptiometry in adults. J Appl Physiol (1985). 2004 Aug;97(2):655-60. doi: 10.1152/japplphysiol.00260.2004. Epub 2004 Apr 16. PMID 15090482
- [Background] Sardinha LB, Lohman TG, Teixeira PJ, Guedes DP, Going SB. Comparison of air displacement plethysmography with dual-energy X-ray absorptiometry and 3 field methods for estimating body composition in middle-aged men. Am J Clin Nutr. 1998 Oct;68(4):786-93. doi: 10.1093/ajcn/68.4.786. PMID 9771855
- [Derived] Nabuco HCG, Tomeleri CM, Fernandes RR, Sugihara Junior P, Venturini D, Barbosa DS, Deminice R, Sardinha LB, Cyrino ES. Effects of pre- or post-exercise whey protein supplementation on oxidative stress and antioxidant enzymes in older women. Scand J Med Sci Sports. 2019 Aug;29(8):1101-1108. doi: 10.1111/sms.13449. Epub 2019 May 27. PMID 31050066
- [Derived] Nabuco HCG, Tomeleri CM, Sugihara P Junior, Fernandes RR, Cavalcante EF, Dos Santos L, Silva AM, Sardinha LB, Cyrino ES. Effect of whey protein supplementation combined with resistance training on cellular health in pre-conditioned older women: A randomized, double-blind, placebo-controlled trial. Arch Gerontol Geriatr. 2019 May-Jun;82:232-237. doi: 10.1016/j.archger.2019.03.007. Epub 2019 Mar 7. PMID 30870778
- [Derived] Nabuco HCG, Tomeleri CM, Sugihara Junior P, Fernandes RR, Cavalcante EF, Venturini D, Barbosa DS, Silva AM, Sardinha LB, Cyrino ES. Effects of pre- or post-exercise whey protein supplementation on body fat and metabolic and inflammatory profile in pre-conditioned older women: A randomized, double-blind, placebo-controlled trial. Nutr Metab Cardiovasc Dis. 2019 Mar;29(3):290-300. doi: 10.1016/j.numecd.2018.11.007. Epub 2018 Nov 29. PMID 30639252
- [Derived] Nabuco HCG, Tomeleri CM, Sugihara Junior P, Fernandes RR, Cavalcante EF, Antunes M, Ribeiro AS, Teixeira DC, Silva AM, Sardinha LB, Cyrino ES. Effects of Whey Protein Supplementation Pre- or Post-Resistance Training on Muscle Mass, Muscular Strength, and Functional Capacity in Pre-Conditioned Older Women: A Randomized Clinical Trial. Nutrients. 2018 May 3;10(5):563. doi: 10.3390/nu10050563. PMID 29751507